CLINICAL TRIAL: NCT04665063
Title: A Multicenter Clinical Study on the Safety and Effectiveness of CAR-T in the Treatment of Relapsed/Refractory Hodgkin's Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020103
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-10

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — CF regimen; Leukapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auto CAR-T (Experimental): Patients will be treated with Auto CAR-T cells
  Interventions: Biological: Auto CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis

INTERVENTIONS:
Biological: Auto CAR-T — Biological: Auto CAR-T
Drug: Cyclophosphamide,Fludarabine — Drug: Cyclophosphamide,Fludarabine
Procedure: Leukapheresis — Leukapheresis

SUMMARY:
This study is a multi-center, non-randomized, single-arm, open clinical trial.

DETAILED DESCRIPTION:
A single car consists of scFv, hinge region, transmembrane region, costimulatory domain and zeta subunit of CD3.Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily sign the informed consent form, and be willing and able to comply with the visits, treatment plans, laboratory inspections, and other requirements of the research as specified in the test procedure;
2. Hodgkin lymphoma patients who are judged to be relapsed/refractory by clinical diagnosis, relapse or refractory are defined as:

   1. Primary resistance to standard treatment regimens;
   2. Or PD occurs after standard treatment with at least second-line standard treatment plan;
   3. Or the last treatment effect is SD and the duration does not exceed 6 months;
   4. Or after anti-PD-1 monoclonal antibody treatment is ineffective or relapses;
   5. Patients who have PD after autologous hematopoietic stem cell transplantation or confirmed recurrence by biopsy within 12 months, or patients who undergo salvage treatment after autologous hematopoietic stem cell transplantation have no remission or relapse after treatment.
3. According to RECIST version 1.1 , there should be at least one measurable tumor;
4. Subjects whose physical status scored by the Eastern Cooperative Oncology Group (ECOG) is 0~2;
5. 14 years old ≤ age ≤ 75 years old, both male and female;
6. Immunohistochemistry or flow cytometry detects tumor cells as CD30 or CD19/CD22/CD79 positive;
7. The estimated survival period from the date of signing the informed consent form is greater than 3 months;
8. Laboratory examinations meet the following conditions: hemoglobin ≥80g/L, platelet count ≥50 × 109/L, absolute neutrophil count (ANC) ≥1.0 × 109/L, if the investigator believes that the above inspection value is below the lower limit It is caused by tumor invading bone marrow and can be included in the group after consultation with the sponsor;
9. The main organ functions need to meet the following conditions: serum creatinine ≤1.5 ULN, AST (aspartate aminotransferase)/ALT (alanine aminotransferase)/ALP (alkaline phosphatase) ≤2.5 ULN, total bilirubin ≤1.5 ULN, left Ventricular ejection fraction (LVEF) ≥50%, and minimum lung function reserve (dyspnea is not higher than level 1 and blood oxygen saturation is greater than 92% under indoor conditions).

Exclusion Criteria:

1. Severe cardiac insufficiency, left ventricular ejection fraction <50%;
2. There is a history of severe lung dysfunction diseases;
3. The patient has had other malignant tumors in the past 5 years, except for skin basal cell carcinoma, breast carcinoma in situ and cervical carcinoma in situ that have undergone radical treatment;
4. Combined with severe or persistent infection and cannot be effectively controlled; Severe infection: Refers to sepsis or uncontrolled infection of the infected foci, and can be included in the group after infection is controlled
5. Combined metabolic diseases (except diabetes);
6. Combined with severe autoimmune disease or innate immune deficiency;
7. Untreated active hepatitis (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] test results are positive, HBV-DNA ≥ 500 IU/ml and abnormal liver function; hepatitis C, defined as hepatitis C antibody [ HCV-Ab] positive, HCV-RNA higher than the detection limit of the analysis method and abnormal liver function) or combined with hepatitis B and C co-infection;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection;
9. A history of severe allergies to biological products (including antibiotics);
10. Participate in any other clinical drug trials at the same time within one month;
11. There are other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the research, or interfere with the results of the research, and patients who the researcher believes are not suitable for participating in this research.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-10-21 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | first one month after CAR-T infusion
  To evaluate the possible adverse events occurred within first one month after CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission (CR), partial remission (PR), objective response (ORR = CR + PR), disease stability (SD), disease progression (PD) and and unresponsive (NR)

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months after CAR-T infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months after CAR-T infusion
  progression-free survival (PFS) time

CONTACTS AND LOCATIONS:
Overall Officials: Baoen Shan, PhD & MD, Principal Investigator — Hebei Medical University Fourth Hospital; Lihong Liu, PhD & MD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Hematology Department, Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China